CLINICAL TRIAL: NCT05883553
Title: Epithesis Versus Prosthesis in Post-phalloplasty Transgender Patients.
Acronym: EROS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: ELATOR/EREKTOR (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ONZ-2023-0121
Record Dates: First submitted 2023-05-09; First posted 2023-06-01 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-08

CONDITIONS: Transgenderism; Erectile Dysfunction; Prosthesis Durability; Gender Dysphoria; Sexual Dysfunction
Keywords: Gender dysphoria; Transgender; Phalloplasty; Erectile dysfunction; Sexual function; Erection prosthesis; Penile epithesis; Medical device; Penile splint; Patient Reported Outcome Measures (PROMs); Genital reconstruction; Reconstructive urology
MeSH Terms: conditions — Transsexualism; Erectile Dysfunction; Prosthesis Failure; Gender Dysphoria; Sexual Dysfunction, Physiological

STUDY DESIGN:
Intervention Model Description: Non-inferiority parallel cohort study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Epithesis group (Experimental): Participants receive an Elator device which was measured to the size of their phallus.
  Interventions: Device: Usability and added value of device within sexual activity
- Prosthesis group (Active Comparator): Participants receive a Zephyr ZSI 475 FTM internal erection prosthesis device as the current standard of care in our hospital. A healing phase of at least six weeks is respected.
  Interventions: Device: Usability and added value of device within sexual activity

INTERVENTIONS:
Device: Usability and added value of device within sexual activity — Participants and there partners will be asked to use the device over the course of 4 months, during which both will provide answers to questionnaires on quality of relation and sexual life, and detailed questions on the usability and the added value of the used device during sexual activity along with overall satisfaction with the device.

SUMMARY:
Transgender and gender diverse (TGD) individuals most often choose for phalloplasty as a means to create masculine external genitalia. The neophallus created in phalloplasty is usually insufficient for penetrative sexual intercourse due to the lack of erectile structures. Therefore, implantation of an internal erectile prosthesis or use of an external device or epithesis is required.

Internal prostheses are the main method for attaining penile rigidity after phalloplasty, but they carry a high risk of complications. Previous research has shown that up to 22% of prostheses for cisgender men were explanted due to various reasons, including infection, erosion, and malfunction within 20 months. The lack of reliable and durable erectile devices leads to a large proportion of patients either choosing phalloplasty but never going for the placement of an erectile prosthesis or completely abandoning the idea of GGAS under the form of phalloplasty. Secondarily, TGD individuals may be concerned about complication rates and likely need for additional surgeries associated with penile implant surgery. Therefore, alternative options for transgender and gender non-conforming patients after phalloplasty are needed. These alternatives may be surgical or non-surgical.

External penile epitheses or penile splints were originally designed for cisgender men with erectile dysfunction but have been used experimentally by post-phalloplasty transgender men. While there is no data on the usability and durability of penile epitheses in a TGD population, they may be a viable alternative to an internal penile prosthesis after phalloplasty. Penile lifters or splints, marketed as ElatorTM or ErektorTM, are commercially available and consist of two rigid rings connected by rigid metal rods. The biggest of two rings is placed around the base of the phallus, and the second ring is placed behind the coronal ridge. By connecting the rods to the ring at the base of the penis, tension and rigidity between the two rings is created, allowing the user to penetrate their partner and remove the device after intercourse.

The current study aims to extend the knowledge on these external devices by comparing them to the implantation of an internal penile prosthesis in post-phalloplasty transgender patients.

DETAILED DESCRIPTION:
Gender dysphoria refers to an inner mental unrest resulting from an incongruity between the assigned biological sex and the mentally experienced sex. The generally accepted treatment for gender dysphoria aims to bring a person's physical characteristics in line with his or her perceived gender identity. This gender-affirming treatment consists of a combination of psychological counselling, hormonal therapy and, if desired, genital gender-affirming surgery (GGAS), which involves the removal of the biological reproductive organs and in some cases (part of) the biological sex organs. These can be replaced by surrogate sex organs of the desired sex while maintaining urological and sexual function. In transgender men, metoidioplasty or phalloplasty are performed. A national survey of transgender adults in the United States has shown that 22% of transgender men have had or clearly state they want gender affirming surgery in the form of phalloplasty, while 27% state this for metoidioplasty. In phalloplasty, anatomically sized external genitalia (penis with or without urethra, scrotum, and perineum) are created using on the one hand a donor skin flap (usually from the forearm, upper leg or inguinal region), and on the other hand tissues from the original genitals. In metoidioplasty, the goal is to create anatomically looking but undersized external genitalia in which the clitoris forms the base of a micro-penis. The neophallus created in the case of phalloplasty is by itself usually insufficient for penetrative sexual intercourse, due to the lack of erectile structures. However, previous research suggests that one of the main reasons transgender male individuals choose for phalloplasty over metoidioplasty is the ability to penetrate a sexual partner. This was also one of the original goals of phalloplasty.

In order to be able to proceed to penetrative sexual intercourse, one option can be the implantation an internal erectile prosthesis or the use of an external device or epithesis. Internal protheses form at this point the main method of attaining penile rigidity after phalloplasty. Both malleable and inflatable options are available today. However, these devices, just as the primary GGAS procedures, carry a high risk of complications. Previous research with prostheses originally designed for cisgender men has shown that up to 22% of prostheses was explanted for various reasons including infection, erosion and malfunction within 20 months. Another study showed that only 62% of patients still had their prosthesis in place after 4 years. More recent publications with a prosthesis specifically designed for phalloplasty patients (ZSITM 475 FtM, Zephyr Surgical Implants, Switzerland, Europe) have shown explantation rates of 19% and 23% at 9 and 18 months respectively. The lack of reliable, and durable erectile devices leads to the fact that a large proportion of patients either chooses for phalloplasty but never goes on the placement of an erectile prothesis or completely abandons the idea of GGAS under the form of phalloplasty at this point in time. As underlined in a recent qualitative study, transgender men may very well be concerned about the complication rates and likely need for additional surgeries associated with the surgical treatments they seek to diminish their gender dysphoria, specifically in penile implant surgery. This is further aggravated by the fact that penile implant surgery is associated with higher complication in a transgender population than in a cisgender population. Penile prostheses were originally designed for an older cisgender male population with treatment resistant erectile disfunction wishing to regain the capacity of penetrative sexual intercourse. No data exists on what the durability of penile implants are in a younger and more sexually active population. Furthermore, the placement of a prosthesis is particularly more difficult after phalloplasty as there are no cavernosal bodies with surrounding tunica albuginea that can be used as scaffold for anchoring of the prosthesis to the pubic bone and preventing it from erosion through the skin. Therefore, alternative options for transgender and gender non-conforming patients after phalloplasty are needed. Although some may be surgical, it may be interesting for some individuals to have non-surgical options as well.

When considering penile epitheses, multiple types are commercially available. One of such devices is a penile lifter or splint and is marketed as the ElatorTM or the ErektorTM for cisgender patients with erectile dysfunction after prostate cancer. These devices consist of two rigid rings connected by rigid metal rods. The biggest of two rings is placed around the base of the phallus. The second ring is connected to the metal rods and is placed behind the coronal ridge. By connecting the rods to the ring at the base of the penis, tension and therefore rigidity between the two rings is created. With the device in place, men can then penetrate their partner and remove it again after intercourse.

Penile splints were originally designed in the beginning of the 20th century for various reasons of erectile disfunction. Loewenstein was the first to produce a study on his personal re-interpretation of this device in 1941. Originally, these devices have been designed for cisgender men with erectile dysfunction, but social media and patient conversations suggest that post-phalloplasty patients have been experimenting with them. Feedback from transgender patients using this device can be found on the website of the product manufacturers, but also on social media sites such as Tumblr, Youtube, and private Facebook channels. They may form a potential alternative to internal prostheses in transgender patients not wishing to undergo further surgery after phalloplasty or in patients that have experienced problems after implantation. A recent study piloting the use of the ElatorTM in 10 post-phalloplasty transgender participants and their partners has suggested that the feasibility of continued use of the epithesis lies around 30%. However, the low patient inclusion rate and substantial loss of follow-up during this preliminary study may very well have biased final results. Nevertheless, important lessons on patients' concerns and expectations as well as anatomical reflections are to be learned from this study. Therefore, our center has been keeping close contact with the team of Dr. Boskey in designing this study protocol.

The current study aims to extend the knowledge on these external devices by comparing them to the implantation of an internal penile prosthesis in post-phalloplasty transgender patients.

ELIGIBILITY:
Inclusion Criteria:

* Transgender or gender non-conforming individuals diagnosed according to the DSM-5 diagnostic criteria for gender dysphoria.
* Patients have undergone phalloplasty as a form of genital gender affirming surgery.
* ≥ 1 year after phalloplasty (any type of flap combination is allowed), performed at the Ghent University Hospital or Amsterdam UMC.
* ≥ 3 months after coronaplasty and having reasonably pronounced coronal ridge, as defined by the surgeons' expert opinion (This criterion is only obligatory in the eptithesis group, not in the prosthesis group).
* Anatomic penile length and girth as defined by the surgeons' expert opinion.
* Absence of urethral stricture or other structural problem resulting in voiding dysfunction.
* Normal uroflowmetry and post-void residue
* Regain of at least minimal protective sensation up to the tip of the phallus as defined by Semmes-Weinstein monofilament testing.
* Established (primary) sexual relationship with partner who is willing to take part in the study.
* Both patient and partner have interest in penetrative sexual intercourse.
* Patient is unable to penetrate the partner (anal or vaginal) adequately sexually without the aid of supportive measures (condom, taping, penile sleeve, penile epithesis or any other measure defined as supportive by the investigators).
* Fit and eligible for erection prosthesis surgery, based on the surgeons' expert opinion.
* No history of erection prosthesis surgery.
* No interest in or fear of prosthesis surgery making this option obsolete (This criterion is only obligatory in the eptithesis group, not in the prosthesis group)
* Treatment naïve in the use of the Elatortm or Erektortm epithesis.
* Voluntarily signed written informed consent according to the rules of Good Clinical Practice (Declaration of Helsinki) and national regulations.

Exclusion Criteria:

* Cisgender patients treated with phalloplasty various reasons.
* Post-metoidioplasty patients (metoidioplasty as step-up to performed phalloplasty is allowed).
* Absence of coronaplasty or coronaplasty performed < 3 months ago or coronaplasty did not leave sufficiently pronounced coronal ridge as defined by the surgeons' expert opinion (This criterion is only obligatory in the epithesis group, not in the prosthesis group)
* Penile dimensions are not anatomic (e.g. too small or too large).
* Underlying LUTDs requiring further investigation and/or treatment.
* Inadequate protective sensation in the penis.
* No established (sexual) partner and/or partner is not willing to take part in the study.
* Patient and/or partner have no interest in penetrative sexual intercourse.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-05-17 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients choosing either for the prosthesis or the epithesis at the start of study | Baseline assessment
  At baseline, patients will get information on both the prosthesis and the epithesis and will be free to choose between them. This difference in percentage and the reasons for choosing between either will be noted.
Difference in capability rate of vaginal and/or anal penetration of the participant's partner | Baseline questionnaire, followed by reassessment at 1 and 4 months after study start
  * Capability will be defined as full repetitive anal and/or vaginal penetration of the partner while using the epithesis or prosthesis, which was not possible before use or implantation, without pain to patient and/or partner, until the end of the intended sexual intercourse.
  * If penetration is not possible, the reasons for this incapacity will be noted

SECONDARY OUTCOMES:
Interest in continued use of epithesis by both patient and partner | Assessment at 4 months after study start
  Interest in continued use will be defined as the proportion of patients and their partners in the epithesis arm with interest in and willingness to continue use of the external penile epithesis after the study period.
Difference in quality of sexual experience | Baseline questionnaire, followed by reassessment shortly after sexual activity. To be filled out by patient and partner at least once per month during the 4 months of the study period
  Assessed using the Quality of Sexual Experience questionnaire (QSE). The QSE questionnaire provides a summative score between 7 and 49. A higher score indicates a better sexual experience.
Difference in treatment satisfaction | Assessment at 1 and 4 months after study start
  Assessed using the Erectile Dysfunction Inventory of Treatment Satisfaction questionnaire (EDITS).
  The EDITS questionnaire provides two summative scores of 0-44 and 0-20 for patient and partner scores respectively. A higher score indicates a better treatment satisfaction. Higher scores indicate better outcome.
Difference in relationship satisfaction | Baseline questionnaire, followed by reassessment at 1 and 4 months after study start
  Assessed using the Maudsley Marital Questionnaire (MMQ). The MMQ provides three summative scores of 0-80, 0-40 and 0-40 on relationship satisfaction, sexual satisfaction, and overall quality of life respectively. Lower scores indicate better outcome.
Difference in lower urinary tract symptoms | Baseline questionnaire, followed by reassessment at 1 and 4 months after study start
  Assessed using the International Consultation on Incontinence Questionnaire Male Lower Urinary Tract Symptoms (ICIQ-MLUTS).
  The ICIQ-MLUTS module, consisting of 7 questions, provides a summative score between 0 (asymptomatic) and 24 (most symptomatic) (question 1 - 6) and a bother score between 0 (not bothersome) and 3 (very bothersome) (question 7).
Difference in maximum flow rate | Baseline evaluation, followed by reassessment at 1 and 4 months after study start
  Assessed using uroflometry (Qmax)
Postoperative complication rate | Within 90 days postoperatively
  Categorized according to Clavien-Dindo classification system
Overall complication rate | Continuously for duration of study period until 90 days after end of study period
  Categorized according to Common Terminology Criteria for Adverse Events classification system (CTCAE)

CONTACTS AND LOCATIONS:
Overall Officials: Nicolaas Lumen, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (2):
- Department of Urology, University Hospital Ghent, Ghent, East-Flanders, Belgium
- Department of Urology, Amsterdam University Medical Center, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No